CLINICAL TRIAL: NCT03605706
Title: A Phase III, Multicentered, Randomized, Double-blinded, Parallel Controlled Study to Evaluate Camrelizumab (PD-1 Antibody) in Combination With FOLFOX4 Regimen Versus Placebo in Combination With FOLFOX4 Regime in First-Line Therapy in Subjects With Advanced Hepatocellular Carcinoma (HCC).
Brief Title: A Trial of SHR-1210 (an Anti-PD-1 Inhibitor) in Combination With FOLFOX4 in Subjects With Advanced HCC Who Have Never Received Prior Systemic Treatment.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1210-III-305-HCC
Record Dates: First submitted 2018-07-22; First posted 2018-07-30 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — camrelizumab; Folfox protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210 (Experimental): SHR-1210+FOLFOX4
  Interventions: Drug: SHR-1210; Drug: FOLFOX4
- CONTROL (Experimental): SHR-1210+Placebo
  Interventions: Drug: FOLFOX4; Drug: Placebo

INTERVENTIONS:
Drug: SHR-1210 — Subjects receive SHR-1210 intravenous at the dose 3mg/kg on Day 1 every 2 weeks
  Arms: SHR-1210
Drug: FOLFOX4 — Subjects receive FOLFOX4 treatment on D1-D2 of every 2 weeks
Drug: Placebo — Subjects receive placebo of SHR-1210 intravenous at the dose 3mg/kg on Day 1 every 2 weeks
  Arms: CONTROL

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR-1210 plus FOLFOX4 in subjects with advanced HCC who have never received prior systemic treatment compared to placebo plus FOLFOX4.

The primary study hyposis is that Camrelizumab combined with FOLFOX4 treatment can improve Overall Survival when compared with placebo in combination with FOLFOX4 Regimen.

ELIGIBILITY:
Inclusion Criteria:

Has not received prior systemic treatment for their advanced/metastatic HCC. Has measurable disease according to RECIST v1.1. ECOG Performance Status of 0 or 1. Child-Pugh Class A or B with 7 points. Life Expectancy of at least 12 weeks. HBV DNA<500 IU/ml. Adequate organ function： Male or female participants of childbearing potential must be willing to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

Known fibrolamellar HCC, Prior malignancy active with the previous 5 years except for locally curable cancers that have been apparently cured.

Known or occurrence of central nervous system (CNS) metastases. Ascites with clinical symptoms. Known or evidence of GI hemorrhage within the past 6 months. Known or occurrence of hemorrhage/ thrombus. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias.

Grade III~IV cardiac insufficiency, according to NYHA criteria or echocardiography check: LVEF<50%.

Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents (systolic blood pressure > 150mmHg, diastolic blood pressure > 90 mmHg).

History of hepatic encephalopathy. Known history of human immunodeficiency virus (HIV) infection. Active infection or an unexplained fever > 38.5°C during screening visits. Prior or planning to organ transplantation including liver transplantation. Interstitial lung disease that is symptomatic or may interfere with the detection and management of suspected drug-related pulmonary toxicity.

Proteinuria≥ 2+ and 24 hours total urine protein > 1.0 g. Active known, or suspected autoimmune disease. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment.

Any loco-regional therapy to liver (included but not limited: resection, radiotherapy, TAE, TACE, TAI, RFA or PEI) within 4 weeks prior to study.

Known history of hypersensitivity to monoclonal antibodies or any components of the study drugs.

Pregnant or breast-feeding women. According to the investigator, other conditions that may lead to stop the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to approximately 3 years
  OS was defined as the time from randomization to death due to any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 in all participants | Up to approximately 6 months
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
Time to Progression (TTP) per RECIST 1.1 in all participants | Up to approximately 3 years
Duration of Response (DoR) per RECIST 1.1 in all participants | Up to approximately 3 years
Disease Control Rate (DCR) per RECIST 1.1 in all participants | Up to approximately 3 years
Progression-free Survival (PFS) per RECIST 1.1 in all participants | Up to approximately 3 years
AE | Up to approximately 3 years
Overall Survival (OS) rate at 9 months and 12 months | Up to approximately 9 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shukui Qing, MD, Study Chair — China, Jiangsu 81 Hospital Nanjing
Locations (1):
- 81 Hospital Nanjing, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No